CLINICAL TRIAL: NCT02281890
Title: Neurodevelopmental Outcomes After Suspected or Proven Sepsis: Secondary Analysis of INIS Trial Database
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: INIS Collaborative Group (Unknown); Maastricht University Medical Center (Other); Erasmus Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: INIS-01
Record Dates: First submitted 2014-10-09; First posted 2014-11-04 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-10

CONDITIONS: Neonatal Sepsis
Keywords: neurodevelopmental disability
MeSH Terms: conditions — Neonatal Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Proven sepsis: Children included in the INIS trial in whom pathogenic organisms (i.e. bacteria or fungi) were cultured from blood and/or cerebrospinal fluid during the sepsis period at the time of study inclusion
  Interventions: Other: Proven sepsis
- Clinical sepsis: Children included in the INIS trial in whom no pathogenic organisms (i.e. bacteria or fungi) were cultured from blood or cerebrospinal fluid during the sepsis period at the time of study inclusion

INTERVENTIONS:
Other: Proven sepsis — Exposure is proven sepsis
  Groups: Proven sepsis

SUMMARY:
Neonatal sepsis is an important determinant of adverse neurodevelopmental outcome. The investigators seek to investigate whether neurodevelopmental outcome following neonatal sepsis differs according to whether or not the diagnosis is confirmed by culture. In a secondary analysis of all 3493 infants included in the International Neonatal Immunotherapy Study (INIS) randomized controlled trial of intravenous immunoglobulin for neonatal sepsis, the investigators will evaluate neurodevelopmental outcomes according to whether or not the sepsis was culture-proven. The primary outcome is death or major disability at two years. In secondary analyses the investigators will determine neurodevelopmental outcomes according to the causative organism identified. Greater understanding of the impact of culture-positivity on long-term outcomes in the setting of clinical neonatal sepsis is essential to better inform parents about the future prospects of their child and to guide patient follow-up.

DETAILED DESCRIPTION:
Rationale Neonatal sepsis is an important determinant of adverse neurodevelopmental outcome [Adams-Chapman 2006, Stoll 2004]. A recent meta-analysis estimated that neonatal sepsis more than doubled the risk of adverse neurodevelopmental outcome in very-low-birth-weight (VLBW) infants (OR 2.09 [95%CI 1.65-2.65]), including cerebral palsy (OR 2.09 [95%CI 1.78-2.45]).[Alshaikh 2013] When a baby with signs suggestive of sepsis, it is common practice to commence intravenous antibiotic treatment as soon as possible after cultures from blood and relevant additional sites have been obtained. However, cultures remain negative in an important subgroup of babies treated for sepsis, despite convincing clinical and/or laboratory signs of sepsis being present. Although there is some evidence to suggest that long-term outcomes following neonatal sepsis may differ according to whether or not the diagnosis was confirmed by culture,[Stoll 2004, Schlapbach 2011] to the best of the investigators' knowledge a direct comparison between these groups has never been made. Greater understanding of the impact of culture-positivity on long-term outcomes in the setting of clinical neonatal sepsis is essential to better inform parents about the future prospects of their child and to guide patient follow-up.

Objective Investigate differences in neurodevelopmental outcome at two years after neonatal sepsis according to whether or not the diagnosis was confirmed by culture.

Research questions Primary Are neurodevelopmental outcomes at two years different between babies with suspected versus culture-proven sepsis? Secondary Are neurodevelopmental outcomes at two years different between babies with suspected versus culture-proven sepsis when considered according to the underlying pathogen?

Design Secondary cohort analysis of all babies included in the International Neonatal Immunotherapy Study (INIS) randomized controlled trial (RCT).[INIS Study Collaborative Group 2008]

Study population The study population consists of all babies included in the INIS trial. The INIS trial was an RCT of intravenous immunoglobulin (two infusions of 500 mg/kg body weight polyvalent IgG) versus placebo in the treatment of suspected or proven neonatal sepsis.[INIS Study Collaborative Group 2008] 3493 infants were included from 113 hospitals in nine countries.[INIS Collaborative Group 2011] There was no difference between the treatment groups in the primary outcome of death or major disability at the age of two years (RR 1.00 [95%CI 0.92-1.08]), or in any of the secondary outcomes. Neither was an effect of immunoglobulin demonstrated in any of the pre-specified subgroup analyses. As the intervention under study did not have an impact on any of the outcomes, secondary observational analyses within the dataset are feasible.

Exposure For the primary analyses two groups of babies with neonatal sepsis will be considered: those with proven sepsis and those with suspected sepsis. Sepsis will be considered proven when pathogenic organisms (i.e. bacteria or fungi) were cultured from blood and/or cerebrospinal fluid. All babies with clinical neonatal sepsis in whom cultures remained negative are considered to have suspected sepsis. In a secondary analysis, neurodevelopmental outcomes of babies with proven sepsis will be compared to those with suspected sepsis according to causative organism grouped as follows: coagulase-negative staphylococci (CONS); other Gram-positive bacteria; Gram-negative bacteria; fungi. Babies will be classified according to the sepsis episode at the time of inclusion in the INIS trail. The impact of any additional episodes of sepsis will be investigated in sensitivity analyses (see below).

Outcomes The primary outcome of interest is death or major disability at two years of age. Secondary outcomes (all at two years of age) include: death; disability; and components of disability: neuromotor disability; disability due to seizures; hearing disability; visual disability; communicative disability; cognitive disability. All types of disability are categorised into major/non-major/no disability. The investigators used two questionnaires; the Health Status Questionnaire (HSQ) was completed by a pediatrician and the Parent Questionnaire (PQ) was completed by a parent or carer. A third questionnaire, the Short Health Status Questionnaire (SHSQ), was developed by the Project Management Group in order to capture the primary outcome for difficult to find children. These questionnaires were sent to general practitioners or health visitors.

The disability classification for each domain (with the exception of the cognitive domain) was calculated from the answers to questions on the HSQ or the PQ [see INIS Collaborative Group 2011 (online supplement) for more detail]. If one questionnaire was missing, the calculation used only the answer on the other questionnaire. If the domain classification was unknown and a SHSQ had been received, the classification from that questionnaire was used for that domain only. Cognitive function was assessed in INIS by parents using the revised Parent Report of Children's Abilities questionnaire (PARCA-R1 [Saudino 1998]), as described previously [INIS Collaborative Group 2011 (online supplement)].

Analyses The following characteristics will be compared between babies with proven and suspected sepsis in tabular form: baseline characteristics, clinical characteristics at presentation with sepsis, neonatal outcome at discharge; outcome at two years. Primary and secondary outcomes at two years will be compared between the two groups in univariable analyses using Chi square test. Multivariable adjustment for potential confounders around birth and at presentation with sepsis (including country and INIS study drug) will be performed using separate logistic regression models for each outcome. The logistic regression models will be considered the primary analyses. Separate models will be constructed for major disability and for any disability (major+non-major).

Subgroup analyses Two sets of subgroup analyses will be undertaken. First, given the difference in aetiology between early onset (<72 hours after birth) sepsis and late onset (>=72 hours after birth) sepsis, the data will be re-analysed according to whether the sepsis episode was early or late onset.

Second, as gestational age is a key determinant of adverse neurodevelopmental outcome, the investigators will undertake a subgroup analysis to investigate the impact of proven versus suspected sepsis on neurodevelopmental outcomes according to whether gestational age at birth was < or ≥ 30 weeks.

Sensitivity analyses Missing values are present for a number of covariates to be included in the multivariable adjustment. By default, logistic regression analysis will be based on babies with complete data only on all variables in the model. The investigators will thus undertake a sensitivity analysis after multiple imputation of missing data on all covariates included in the primary model, creating and analysing five unique datasets.

For the primary analysis of this study, only the neonatal sepsis episode at presentation (i.e. at inclusion in the INIS trial) will be considered to classify babies as having suspected or proven sepsis. An important subgroup of babies however, experienced one or more additional episodes of sepsis following inclusion in the study, which may affect the findings depending on whether or not these were culture-proven. The investigators will therefore undertake two additional sensitivity analyses to assess the impact of subsequent episodes of sepsis on the difference in neurodevelopmental outcome according to whether or not proven sepsis was present. In a first sensitivity analysis the investigators will exclude from the cohort all babies in whom additional episodes of neonatal sepsis were present following the initial presentation with sepsis. This will facilitate a fair comparison of babies with single episodes of proven versus suspected sepsis. In a second sensitivity analysis of the full cohort, the investigators will re-classify as proven sepsis all babies labeled as suspected sepsis based on the initial presentation, in whom subsequent episodes of proven sepsis were present. The investigators will then compare neurodevelopmental outcomes according to whether or not proven sepsis was present at any time point during initial hospital admission.

Sample size The sample size of the cohort is based on the original RCT design.[INIS Study Collaborative Group 2008, INIS Collaborative Group 2011] For the purpose of this secondary analysis the cohort may thus be considered a convenience sample. To the best of the investigators' knowledge this cohort is the second largest to evaluate neurodevelopmental outcomes following neonatal sepsis.[Alshaikh 2013] In multivariate analyses of 6093 extremely-low-birth-weight (ELBW) infants from the National Institute of Child Health and Human Development (NICHD) cohort followed up at two years of age, Stoll and colleagues were able to demonstrate clinically relevant differences (OR ≥1.3) in key neurodevelopmental outcomes between uninfected babies and different categories of babies with neonatal sepsis with statistical significance.[Stoll 2004] The same accounted for their subgroup analyses according to causative organism.[Stoll 2004] In much smaller studies, others have also demonstrated statistically significant impact of neonatal sepsis on neurodevelopmental outcome, as reviewed elsewhere.[Alshaikh 2013] The investigators therefore expect the INIS cohort to have sufficient power to detect clinically relevant differences (OR ≥1.3) in neurodevelopmental outcomes between VLBW infants with suspected versus proven neonatal sepsis.

Ethical considerations The original RCT was approved by the national and local ethical committees of each participating hospital. Anonymised data were used for the purpose of this secondary analysis. According to UK and Dutch regulations, no formal ethical assessment is required for secondary analyses of anonymised data.

Dissemination Findings will be reported in a manuscript to be submitted for publication with a leading medical journal in an appropriate field (i.e. paediatrics, infection/immunology, neurology), and may be presented at international clinical and research meetings.

ELIGIBILITY:
Inclusion Criteria:

* Children included in the INIS trial

Exclusion Criteria:

* None

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population consists of all babies included in the INIS trial. The INIS trial was an RCT of intravenous immunoglobulin (two infusions of 500 mg/kg body weight polyvalent IgG) versus placebo in the treatment of suspected or proven neonatal sepsis.[5] 3493 infants were included from 113 hospitals in nine countries.[6]
Sampling Method: Non-Probability Sample
Enrollment: 3493 (Actual)
Dates: Start 2001-10; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
death or major disability | 2 years
  Death or major disability at two years of age. The diagnosis of major disability was based on the answers to questions on the HSQ or the PQ [see Study Description and INIS Collaborative Group 2011 (online supplement) for more detail]. If the domain classification was unknown and a SHSQ had been received, the classification from that questionnaire was used for that domain only.

SECONDARY OUTCOMES:
death | two years
  death before two years of age
disability | two years
  Disability at two years of age, categorised as major or non-major. The diagnosis of disability was based on the answers to questions on the HSQ or the PQ [see Study Description and INIS Collaborative Group 2011 (online supplement) for more detail]. If the domain classification was unknown and a SHSQ had been received, the classification from that questionnaire was used for that domain only.
disability due to seizures | two years
  Disability due to seizures at two years of age, categorised as major or non-major. The diagnosis of disability due to seizures was based on the answers to questions on the HSQ or the PQ [see Study Description and INIS Collaborative Group 2011 (online supplement) for more detail]. If the domain classification was unknown and a SHSQ had been received, the classification from that questionnaire was used.
hearing disability | two years
  Hearing disability at two years of age, categorised as major or non-major. The diagnosis of hearing disability was based on the answers to questions on the HSQ or the PQ [see Study Description and INIS Collaborative Group 2011 (online supplement) for more detail]. If the domain classification was unknown and a SHSQ had been received, the classification from that questionnaire was used.
visual disability | two years
  Visual disability at two years of age, categorised as major or non-major. The diagnosis of visual disability was based on the answers to questions on the HSQ or the PQ [see Study Description and INIS Collaborative Group 2011 (online supplement) for more detail]. If the domain classification was unknown and a SHSQ had been received, the classification from that questionnaire was used.
communicative disability | two years
  Communicative disability at two years of age, categorised as major or non-major. The diagnosis of communicative disability was based on the answers to questions on the HSQ or the PQ [see Study Description and INIS Collaborative Group 2011 (online supplement) for more detail]. If the domain classification was unknown and a SHSQ had been received, the classification from that questionnaire was used.
cognitive disability | two years
  Cognitive disability at two years of age, categorised as major or non-major. The diagnosis of cognitive disability was based on PARCA-R1 [Saudino 1998], as described previously [INIS Collaborative Group 2011 (online supplement)]
neuromotor disability | two years
  Neuromotor disability at two years of age, categorised as major or non-major. The diagnosis of neuromotor disability was based on the answers to questions on the HSQ or the PQ [see Study Description and INIS Collaborative Group 2011 (online supplement) for more detail]. If the domain classification was unknown and a SHSQ had been received, the classification from that questionnaire was used.

CONTACTS AND LOCATIONS:
Overall Officials: Ben Stenson, MD, Principal Investigator — University of Edinburgh; Peter Brocklehurst, MD, Principal Investigator — University of Oxford

REFERENCES:
- [Background] Adams-Chapman I, Stoll BJ. Neonatal infection and long-term neurodevelopmental outcome in the preterm infant. Curr Opin Infect Dis. 2006 Jun;19(3):290-7. doi: 10.1097/01.qco.0000224825.57976.87. PMID 16645492
- [Background] Stoll BJ, Hansen NI, Adams-Chapman I, Fanaroff AA, Hintz SR, Vohr B, Higgins RD; National Institute of Child Health and Human Development Neonatal Research Network. Neurodevelopmental and growth impairment among extremely low-birth-weight infants with neonatal infection. JAMA. 2004 Nov 17;292(19):2357-65. doi: 10.1001/jama.292.19.2357. PMID 15547163
- [Background] Alshaikh B, Yusuf K, Sauve R. Neurodevelopmental outcomes of very low birth weight infants with neonatal sepsis: systematic review and meta-analysis. J Perinatol. 2013 Jul;33(7):558-64. doi: 10.1038/jp.2012.167. Epub 2013 Jan 17. PMID 23328927
- [Background] Schlapbach LJ, Aebischer M, Adams M, Natalucci G, Bonhoeffer J, Latzin P, Nelle M, Bucher HU, Latal B; Swiss Neonatal Network and Follow-Up Group. Impact of sepsis on neurodevelopmental outcome in a Swiss National Cohort of extremely premature infants. Pediatrics. 2011 Aug;128(2):e348-57. doi: 10.1542/peds.2010-3338. Epub 2011 Jul 18. PMID 21768312
- [Background] INIS Study Collaborative Group. The INIS Study. International Neonatal Immunotherapy Study: non-specific intravenous immunoglobulin therapy for suspected or proven neonatal sepsis: an international, placebo controlled, multicentre randomised trial. BMC Pregnancy Childbirth. 2008 Dec 8;8:52. doi: 10.1186/1471-2393-8-52. PMID 19063731
- [Background] INIS Collaborative Group; Brocklehurst P, Farrell B, King A, Juszczak E, Darlow B, Haque K, Salt A, Stenson B, Tarnow-Mordi W. Treatment of neonatal sepsis with intravenous immune globulin. N Engl J Med. 2011 Sep 29;365(13):1201-11. doi: 10.1056/NEJMoa1100441. PMID 21962214
- [Background] Saudino KJ, Dale PS, Oliver B, Petrill SA, Richardson V, Rutter M, Simonoff E, Stevenson J, Plomin R. The validity of parent-based assessment of the cognitive abilities of two-year olds. British Journal of Developmental Psychology 16: 349-363, 1998.